CLINICAL TRIAL: NCT05477667
Title: Study of Let-7a and miRNA-124 in Cases of Non-Hodgkin's Lymphoma and Acute Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Talal Mahmoud, assisstent professor at clinical pathology department at faculty of medicine sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-22-7-22
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Non Hodgkin Lymphoma and Acute Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): the patients with non-malignant hematological diseases
  Interventions: Diagnostic Test: real time pcr
- the cases (A) (Active Comparator): NHL .
  Interventions: Diagnostic Test: real time pcr
- the cases (B) (Active Comparator): acute leukemia
  Interventions: Diagnostic Test: real time pcr

INTERVENTIONS:
Diagnostic Test: real time pcr — Detection of expressin level of MiRNA-124 and let-7a using real time pcr

SUMMARY:
MiRNAs are noncoding RNAs (ncRNAs) that drive post-transcriptional negative regulation of gene expression by promoting the degradation or translational blockade of their target mRNAs. MiRNAs are 21-24-nucleotide-long RNA molecules that are processed from longer RNA precursors (pri-miRNAs) , and either the 5' or the 3' strand of the mature miRNA duplex is loaded into the Argonaute (AGO) family of proteins to form a miRNA-induced silencing complex (miRISC) When bound to AGO proteins, mature miRNAs destabilize or inhibit the translation of partially complementary target mRNAsMiRNA-124 has been shown to be a tumor suppressor, and a decrease in its expression level is typical of tumors of various localization, but there is no evidence of the role of miRNA-124 in the development of NHL . There are a number of studies reflecting the involvement of miRNA-124 in hematopoiesis. Liu et al. showed that miRNA-124 regulates Tip110 that is involved in the differentiation of hematopoietic stem cellsThe let-7 family has been shown to influence the pathogenesis of a variety of hematological malignancies through the changing expression of a number of oncogenic pathways, particularly those related with MYC and that might affect hematopoietic carcinogenesis through the modulation of inflammatory pathways

ELIGIBILITY:
Inclusion Criteria:

* approval to sign an informed written consent,
* patient with NHL and acute leukemia .

Exclusion Criteria:

* Refusal to sign an informed written consent,
* patient on chemotherapy

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
MiRNA-124 level | 6 months
  Detection of expressin level of MiRNA-124 IN Non-Hodgkin's Lymphoma and acute leukemia
let-7a level | 6 months
  Detection of expressin level of let-7a IN Non-Hodgkin's Lymphoma and acute leukemia

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Armitage JO, Gascoyne RD, Lunning MA, Cavalli F. Non-Hodgkin lymphoma. Lancet. 2017 Jul 15;390(10091):298-310. doi: 10.1016/S0140-6736(16)32407-2. Epub 2017 Jan 31. PMID 28153383
- [Background] Bedewy AML, Elmaghraby SM, Shehata AA, Kandil NS. Prognostic Value of miRNA-155 Expression in B-Cell Non-Hodgkin Lymphoma. Turk J Haematol. 2017 Aug 2;34(3):207-212. doi: 10.4274/tjh.2016.0286. Epub 2017 Feb 1. PMID 28148469
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Fuertes T, Ramiro AR, de Yebenes VG. miRNA-Based Therapies in B Cell Non-Hodgkin Lymphoma. Trends Immunol. 2020 Oct;41(10):932-947. doi: 10.1016/j.it.2020.08.006. Epub 2020 Sep 1. PMID 32888820